CLINICAL TRIAL: NCT06582160
Title: Enhancing Uptake of Preconception Care Services in Family Practice Clinics Using a Patient Centered Screening Tool: A Pilot Study
Brief Title: Enhancing Uptake of Preconception Care Services in Family Practice Clinics Using a Patient Centered Screening Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0422-22-EP
Record Dates: First submitted 2024-08-26; First posted 2024-09-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Women; Reproductive Age

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of three conditions upon enrollment: 1) Long form screening; 2) Short form screening; 3) control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient-centered Pre-conception Screening (Experimental): A short form, 2 question screening form which asks participants which preconception health topics they would like to discuss with their doctor today. Includes an option for "None of these. I would not like to discuss how my health can affect fertility and any future pregnancies"
  Interventions: Other: Patient-centered Pre-conception Screening
- Risk-based Pre-conception Screening (Active Comparator): A long form questionnaire screening for a range of preconception health risk factors including: age, weight, exercise, diet, nutrition, health conditions, risky behaviors, immunization status, prescription medications, birth control use
  Interventions: Other: Risk-Based Pre-conception Screening
- Control (No Intervention): Participant is asked a single question: "Your health today can make a difference for the pregnancy you experience tomorrow. Do you agree with the statement above?"

INTERVENTIONS:
Other: Risk-Based Pre-conception Screening — A long form questionnaire screening questionnaire administered via tablet in health clinic waiting room. Offered to participants when checking-in for appointment.
  Arms: Risk-based Pre-conception Screening
Other: Patient-centered Pre-conception Screening — A short form, 2 question screening administered via tablet in health clinic waiting room. Offered to participants when checking-in for appointment.
  Arms: Patient-centered Pre-conception Screening

SUMMARY:
Sixteen years have passed since the Centers for Disease Control recommended routine preconception screening and counseling in primary care settings, yet time constraints and low preconception counseling adherence have prevented widespread uptake. This innovative, self-selected preconception screening tool encourages participants to be active in their own care and eliminates the time burden associated with typical pre-selected screening in clinics. This project will generate important knowledge about the promise of utilizing a participant-selected preconception screening tool to promote preconception health behavior change during routine medical encounters for women of reproductive age.

DETAILED DESCRIPTION:
Women who make positive health behavior changes to protect their fetus typically do so after learning about the pregnancy, unaware that the period of maximum sensitivity to these changes has passed. Fewer than half of mothers enter pregnancy at a healthy weight and an increasing percentage of pregnancies are affected by chronic hypertension and other chronic health conditions. These risk factors are predictive of poor birth outcomes and increased risk to maternal health, yet they are difficult to modify after conception. Routine pre-onception screening and counseling is recommended for all women of reproductive age, yet adherence is low. More than sixteen years after the Centers for Disease Control (CDC) recommended routine preconception screening and counseling in primary care settings, fewer than one-fifth of primary care providers conduct this critical screening. Pioneering approaches are needed to increase preconception screening and improve patient adherence to preconception recommendations in primary care settings. This innovative, self-selected preconception screening tool encourages patients to be active participants in their own care and eliminates the time burden associated with typical pre-selected screening. Typical pre-selected risk screening tools ask patients a series of predetermined health-related questions to identify health risks. Pre-selected tools identify health information needs for the participant, based on the participant's response to the risk assessment. This study proposes a patient-selected screening tool, whereby the participant selects from a list of preconception counseling topics based on her own perceived need for information. This tool has fewer questions, reducing time burden. The first specific aim of this project is to compare topics identified for counseling and overall identification of risk between the two screening approaches. The second aim is to compare preconception knowledge, behavior change intention and self-efficacy between participant who receive participant-selected and pre-selected preconception screening. The third aim is to utilize a QUAN-qual sequential mixed methods design to explain quantitative results and identify novel options for preconception counseling. To accomplish this objective, a pilot study will be conduct in a mid-size primary care clinic located in a Midwest urban setting. Female participants of child-bearing age will be randomly assigned to receive: 1) pre-selected preconception screening; 2) participant-selected preconception risk screening; or 3) no screening. Participants will then be invited to a follow-up interview. Participants will be asked about their experiences with the preconception tools and how to better incorporate preconception screening and counseling into primary care settings. The findings from the quantitative pilot study will be integrated with the qualitative data using an explanatory sequential joint display. This project's results can demonstrate the relevance of utilizing a quicker and potentially more effective preconception screening tool for improving maternal and child health.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female
* Child-bearing age
* Visiting the clinic for a routine or preventative appointment during the study period

Exclusion Criteria:

* Under 19 or over 49 years of age
* Not biologically female

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 286 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Risk Detection Rate | 18 month duration of study
  Percentage of participants identified as having at least one preconception risk factor. Risk rate will be compared between the two types of screen tool (Group 1 - Short Form/Patient Centered and Group 2 - Long Form/Risk Based). Risk detection rates between the two screening methods will be compared against the benchmark risk as assessed in the post-visit questionnaire.
Screening Tool Completion Rate | 18 month duration of study
  Rate of completion for each screening tool. Percent of participants with 75% completion of the screening tool will be compared across Group 1 (Short Form/Patient Centered) and Group 2 (Long Form/Risk Based).
Health Care Relationship Trust Scale - Revised | 18 month duration of the study
  Participants trust in their health care provider will be measured using the Health Care Relationship Trust Scale - Revised (HCR Trust Scale-R). HCR Trust Scale-R scores range from 0 to 52, which higher scores indicating greater levels of trust. The instrument will be administered in the post-visit questionnaire. Trust scores will be compared across intervention arms and against the control group.
Preconception Health Behavior Intentions | 18 month duration of the study
  Intention to change health behavior and self-efficacy for change in response to identified health risks. Measured in the post-visit questionnaire, through the Patient Enablement Instrument (PEI). PEI scores range from 0 to 12, which higher scores indicating greater levels of patient enablement. Additionally, the research team developed two survey items. One item asks respondents if they have the knowledge and skills to improve their preconception health. Response options are yes or no. The second item asks how confident respondents feel that they will make at least one preconception health change. Response options follow Likert scale (1-4) ranging from "Not at all confident" to "Extremely confident." Comparisons in preconception health behavior intention will be compared between both intervention arms, and against the control group.
Preconception Knowledge | 18 month duration of the study
  Awareness of basic preconception health care was assessed through the post-visit questionnaire. To assess knowledge, participants read the following statement: "The following are a set of statements about health and pregnancy. Please answer whether you agree, disagree or are unsure about these statements." This was followed by a series of statements about preconception health such as: "Folic acid should be taken before pregnancy;" "A person's weight when they become pregnant can affect the pregnancy; and "Certain health conditions, like diabetes and hypertension can increase the chances of pregnancy complications." Possible responses were "Agree," "Disagree," or "Unsure." Scores range from 0 to 10, with higher scores indicated higher knowledge. Preconception awareness will be compared across the two intervention groups and against the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon I Maloney, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Nebraska Medicine - Fontenelle Clinic, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No